CLINICAL TRIAL: NCT07171112
Title: Smoking Cessation Treatment Escalation Among Patients With Recurrent Acute Pancreatitis and Chronic Pancreatitis
Brief Title: Smoking Cessation Trial in Recurrent Acute Pancreatitis and Chronic Pancreatitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Samuel Han, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 25-004013
Record Dates: First submitted 2025-08-29; First posted 2025-09-12 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Pancreatitis, Chronic; Pancreatitis, Acute; Recurrent Acute Pancreatitis; Smoking (Tobacco) Addiction
Keywords: Smoking cessation; chronic pancreatitis; recurrent acute pancreatitis; varenicline; bupropion
MeSH Terms: conditions — Pancreatitis, Chronic; Pancreatitis; Smoking; Behavior, Addictive; Smoking Cessation | interventions — BID protein, human; Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Continuation of standard varenicline dosing (1mg BID) (Active Comparator): 1. A group that continues to take varenicline 1mg twice a day (no change)
  Interventions: Drug: Standard Varenicline Dosing (1 mg BID)
- Combination Therapy of varenicline 1mg BID with the addition of bupropion 150 mg BID (Experimental): A group assigned to the combination of standard varenicline dosing (1 mg PO BID) with bupropion (150 mg PO BID)
  Interventions: Drug: Standard Varenicline Dosing (1 mg BID); Drug: Bupropion 150 mg twice daily
- Increased Varenicline Dosing (1 mg TID) (Experimental): A group assigned to increased varenicline (1mg oral three times a day) dosing
  Interventions: Drug: Increased Varenicline Dosing (1mg TID)

INTERVENTIONS:
Drug: Standard Varenicline Dosing (1 mg BID) — Varenicline PO (oral) 1mg twice daily
  Arms: Combination Therapy of varenicline 1mg BID with the addition of bupropion 150 mg BID; Continuation of standard varenicline dosing (1mg BID)
Drug: Bupropion 150 mg twice daily — Bupropion 150 mg PO twice daily
  Arms: Combination Therapy of varenicline 1mg BID with the addition of bupropion 150 mg BID
Drug: Increased Varenicline Dosing (1mg TID) — Varenicline 1mg PO (oral) three times daily
  Arms: Increased Varenicline Dosing (1 mg TID)

SUMMARY:
The purpose of this research is to assess the effectiveness of two treatment strategies for smoking cessation in patients with acute recurrent pancreatitis or chronic pancreatitis who smoke cigarettes. All participants will receive varenicline, a commonly used medication that helps people stop smoking, at its standard dose. For those who are unable to stop smoking after 6 weeks of treatment, they will be randomly selected to either 1) increase their dose of varenicline, 2) combine varenicline with bupropion (another medication that helps with smoking cessation) or continue on the standard dose of varenicline. At the end of 12 weeks of treatment, participants will be asked if they have stopped smoking with confirmation done by measuring carbon monoxide levels in their breath.

DETAILED DESCRIPTION:
This randomized trial evaluates the safety and efficacy of varenicline-based smoking cessation treatment for patients with recurrent acute pancreatitis and chronic pancreatitis. Participants who currently smoke cigarettes and have a desire to quit smoking will be eligible to participate in this study.

Upon providing informed consent, baseline information regarding quality of life, pain, smoking history, and mental health will be collected for each participant in addition to an exhaled carbon monoxide level measurement. Participants will then be started on standard varenicline dosing for smoking cessation (1mg PO BID) for 6 weeks. Participants who continue to smoke (non-abstainers) after 6 weeks will then be randomized into 3 treatment options:

1) Increased varenicline dosing (1mg PO TID) 2) Combination of varenicline (1mg PO BID) with bupropion (150mg PO BID) or 3) Continued standard dosing of varenicline (1 mg PO BID) for an additional 6 weeks.

After 12 weeks of treatment, participants will be asked about their smoking status, have an exhaled carbon monoxide level measured and will repeat their assessments of quality of life, pain, mental health and smoking urges.

ELIGIBILITY:
Inclusion Criteria

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 18 or older
* Diagnosed with either recurrent acute pancreatitis or chronic pancreatitis as defined by the American Pancreatic Association:

  o Chronic Pancreatitis (any of the following): i. Moderate/marked pancreas imaging morphology (i.e. ductal and parenchymal abnormalities ii. Pancreatic calcifications iii. Histologic confirmation

  o Recurrent Acute Pancreatitis: i. Two or more documented attacks of acute pancreatitis, separated by 3 months from one another, defined by at least 2 of the following 3:
  1. amylase or lipase values, or both, that are greater than 3 times the upper limit of normal values
  2. characteristic cross-sectional imaging
  3. typically upper abdominal pain according to the revised Atlanta classification
* Currently smoking ≥ 5 cigarettes/day
* Explicitly express a desire to quit within 30 days
* Ability to take oral medication and be willing to adhere to the study intervention regimen
* Willing and able to comply with trial protocol and follow-up

Exclusion Criteria

* Age < 18 years
* Ongoing acute pancreatitis or prior episode of pancreatitis in previous 30 days
* No desire to quit smoking
* Currently undergoing smoking cessation intervention (i.e. nicotine replacement therapy, varenicline, counseling, bupropion).
* Known allergic reactions to varenicline or bupropion SR
* History of seizures
* History of an eating disorder (anorexia or bulimia)
* Closed head trauma with any loss of consciousness or amnesia in the last 5 year
* Ever history of closed head trauma with > 30 minutes of loss of consciousness or amnesia or resulting in skull fracture or subdural hematoma/brain contusion
* Ever history of alcohol withdrawal
* Ever history of chronic kidney disease (creatine clearance < 30 mL/minute)
* Liver impairment (i.e. history of cirrhosis) with aminotransferase elevation ≥ 2 times the upper limit of normal and/or alkaline phosphatase elevation ≥ 2 times the upper limit of normal.
* History of bipolar disorder or psychosis
* Ongoing or recent use (prior 14 days) of any monoamine oxidase inhibitors (isocarboxazid, phenelzine, tranylcypromine, selegiline).
* Regular use of potent CYP2B6 inhibitors (i.e. clopidogrel, ticlopidine)
* Regular use of CYP2D6 substrates with narrow therapeutic indices (e.g. flecainide, propafenone, tricyclic antidepressants such as nortriptyline, thioridazine, vinblastine)
* History of acute angle closure glaucoma
* Meet criteria for depression as assessed by the Center for Epidemiologic Studies - Depression (CES-D) with a score of 16 or higher.
* Psychiatric hospitalization within 1 year of screening
* Participants who have a score of 3 or higher on the Columbus-Suicide Severity Rating Scale (C-SSRS) at enrollment or during any of the study assessments will be excluded
* Unable to provide consent for self Incarcerated
* Pregnant females. All female patients of childbearing potential must have a negative pregnancy test and must agree to use highly effective (failure rate <1%) contraception during participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who quit smoking at 12 weeks of treatment | 12 weeks
  This outcome measures the number of participants who quit smoking (out of the total number of participants for that intervention arm) after 12 weeks of treatment. Smoking cessation is assessed using a questionnaire that directly asks participants if they have smoked any cigarettes in the last 7 days. Smoking cessation is then confirmed by measuring an exhaled carbon monoxide level using a carbon monoxide monitor.

SECONDARY OUTCOMES:
Proportion of participants who have quit smoking 24 weeks after treatment initiation | 24 weeks
  This outcome measures the number of participants who have quit smoking (out of the total number of participants for that intervention arm) 24 weeks after starting treatment. Smoking cessation is assessed using a questionnaire that directly asks participants if they have smoked any cigarettes in the last 7 days.
Reduction in Smoking | 12 weeks and 24 weeks
  Number of cigarettes smoked per day. This outcome measures whether there has been any change (decrease) in the number of cigarettes smoked a day.
Serious quit attempts | 12 weeks
  Number of attempts where smoking was stopped for at least 24 hours. This outcome measures the number of quitting attempts made by participants during the 12 weeks of treatment.
Treatment Engagement and Retention | 12 weeks
  What proportion of participants adhered to the study protocol and continued with the study until completion
Treatment Acceptability | 12 weeks
  This outcome measures whether the assigned treatment was acceptable to participants. This will be assessed using the Treatment Evaluation Inventory - Short Form (score range 9-45, with higher scores representing greater acceptance of the treatment). This questionnaire uses a 5-point scale and contains 9 questions. A total score of 27 or higher would demonstrate moderate treatment acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Han, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data including participant and disease characteristics and treatment outcomes will be shared.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 24 months after publication of primary manuscript to 5 years after publication of primary manuscript.
Access Criteria: Researchers will be able to access the IPD after submitting a proposal that is reviewed and approved by the PI.
  Deidentified data in accordance to the agreed-upon proposal will be made available to researchers.

REFERENCES:
- [Background] Ebbert JO, Hatsukami DK, Croghan IT, Schroeder DR, Allen SS, Hays JT, Hurt RD. Combination varenicline and bupropion SR for tobacco-dependence treatment in cigarette smokers: a randomized trial. JAMA. 2014 Jan 8;311(2):155-63. doi: 10.1001/jama.2013.283185. PMID 24399554
- [Background] Cinciripini PM, Green CE, Shete S, Minnix JA, Robinson JD, Cui Y, Kim S, Kypriotakis G, Beneventi D, Blalock JA, Versace F, Karam-Hage M. Smoking Cessation After Initial Treatment Failure With Varenicline or Nicotine Replacement: A Randomized Clinical Trial. JAMA. 2024 May 28;331(20):1722-1731. doi: 10.1001/jama.2024.4183. PMID 38696203